CLINICAL TRIAL: NCT04547166
Title: A Randomized, Double-blind, Multicenter, PhaseⅡ/Ⅲ Clinical Study of Serplulimab in Combination With Bevacizumab and Chemotherapy (XELOX) Versus Placebo in Combination With Bevacizumab and Chemotherapy (XELOX) in First-line Treatment of Patients With Metastatic Colorectal Cancer (mCRC)
Brief Title: A Clinical Study to Evaluate Efficacy and Safety of Serplulimab（HLX10） Combined With Bevacizumab（HLX04) and Chemotherapy (XELOX) in Patients With Metastatic Colorectal Cancer (mCRC)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shanghai Henlius Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HLX10-015-CRC301
Record Dates: First submitted 2020-09-07; First posted 2020-09-14 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Serplulima +Bevacizumab+XELOX (Experimental): Serplulimab (HLX10) in Combination With Bevacizumab and chemotherapy (XELOX)
  Interventions: Drug: HLX10; Drug: HLX04、
- placebo + Bevacizumab+XELOX (Placebo Comparator): placebo in combination with Bevacizumab and chemotherapy (XELOX)
  Interventions: Drug: HLX04、

INTERVENTIONS:
Drug: HLX10 — a single fixed dose of 300 mg, intravenous infusion (IV), every 3 weeks (Day 1 of each cycle [D1]), non-reducible.
  Other Names: serplulimab
  Arms: Serplulima +Bevacizumab+XELOX
Drug: HLX04、 — 7.5mg/kg, IV, every 3 weeks (D1 of each cycle), non-reducible.
  Other Names: Bevacizumab

SUMMARY:
This is a two-arm, randomized, double-blinded, multicenter phase III clinical study to evaluate the clinical efficacy of Serplulimab (HLX10) in Combination With Bevacizumab and Chemotherapy (XELOX) Versus Placebo in Combination With Bevacizumab and Chemotherapy (XELOX) in First-line Treatment of Patients With Metastatic Colorectal Cancer (mCRC)

DETAILED DESCRIPTION:
Patients with confirmed unresectable metastatic/recurrent colorectal adenocarcinoma who have not received systemic anti-neoplastic therapy for metastatic/recurrent lesions will be included in this study.Approximately 6-12 patients will be enrolled in the Part I (Safety Run-in Period).Approximately 100 patients will be enrolled in the Part II (Phase II study, 50 in the test group and 50 in the control group).Approximately 568 patients will be enrolled in the Part III (Phase III study, 284 in the test group and 284 in the control group).

Part II (Phase II study): Approximately 40 study sites in China will participate.

Part III (Phase III study): A total of approximately 75 study sites in 3 countries(including China, Japan, Indonesia) will participate.

The study consists of a screening period (up to 28 days), a treatment period (3-week cycle, up to 2 years), and a follow-up period (including a safety follow-up period, and a survival follow-up every 12 weeks).

ELIGIBILITY:
Key Inclusion Criteria:

1. Histopathologically confirmed unresectable metastatic/recurrent colorectal adenocarcinoma
2. Life expectancy ≥ 12 weeks
3. Have not received any previous systemic anti-tumor drug treatment for metastatic colorectal adenocarcinoma
4. For participants who have previously received neoadjuvant/adjuvant therapy, the time from the last treatment to recurrence or progression must exceed 12 months.
5. With at least one measurable lesion as assessed by the IRRC per RECIST v1.1, and the measurable lesion should not have been treated locally such as with radiotherapy (a lesion located in an area subjected to previous radiotherapy can also be regarded as a measurable lesion if PD is confirmed)
6. Agree to provide sufficient previously preserved tumor tissue specimens or agree to undergo biopsy to collect tumor tissue for some gene test.
7. Have an ECOG PS score of 0 or 1 within 7 days prior to receiving the first dose of the study drugs
8. Have Adequate major organ functions.

Key Exclusion Criteria:

1. Have confirmed MSI-H CRC (gene test)
2. Subjects with oligometastatic liver disease and presenting the potential for becoming resectable
3. Presence of central nervous system (CNS) or leptomeningeal metastases
4. Have received radiotherapy within 6 months prior to the initiation of study treatment, except for palliative radiotherapy for bone disorders at least 14 days prior to initiation of study treatment; radiotherapy covering more than 30% of the bone marrow area within 28 days prior to randomization is not allowed.
5. With a history of or current interstitial pneumonia, pneumoconiosis, radiation pneumonitis, drug-related pneumonitis, severe pulmonary dysfunction, or any condition that may interfere with the detection and management of suspected drug-related pulmonary toxicity
6. Have received major surgery within 28 days prior to randomization. A major surgery in this study is defined as a surgery requiring at least 3 weeks of recovery to be able to receive the treatment in this study
7. Previously received intestinal stent implantation, with the stent remaining in place at the screening period
8. Uncontrolled hypertension despite clinical treatment (defined as systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 100 mmHg)
9. With a history of hypertensive crisis or hypertensive encephalopathy
10. With a history of significant/severe hemorrhage within 1 month prior to randomization, or have received blood transfusion within 2 weeks prior to randomization
11. Requiring long-term treatment with daily administration of nonsteroidal anti-inflammatory drugs (NSAIDs). Occasional use of NSAIDs to relieve medical symptoms such as headache or pyrexia is allowed
12. With evidence showing the presence of meteorism that cannot be attributed to puncture or recent surgery
13. Presence of severe, unhealed or split wounds and active ulcers or untreated fractures
14. Presence of any of the following medical conditions within 6 months prior to randomization:

    1. Abdominal or tracheoesophageal fistula, gastrointestinal perforation or intra-abdominal abscess, massive ascites as judged by the investigator (defined as patients requiring drainage or treatment within two weeks)
    2. Intestinal obstruction and/or previous clinical signs or symptoms of gastrointestinal obstruction, including incomplete obstruction associated with a preexisting disease or requiring routine parenteral hydration, parenteral nutrition, or tube feeding. 2 months prior to randomization, patients with previous symptoms of incomplete obstruction/obstructive syndrome/signs/symptoms of intestinal obstruction that have improved after treatment may be enrolled in the study as assessed by the investigator
    3. Severe, uncontrollable intra-abdominal inflammation requiring clinical intervention as judged by the investigator
    4. Major vascular disease (e.g., aortic aneurysm requiring surgical repair or associated with recent peripheral artery thrombosis)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 568 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2025-09-24 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival (assessed by independent radiological review committee (IRRC) based on RECIST v1.1)

SECONDARY OUTCOMES:
OS | From date of randomization until the date of first date of death from any cause, assessed up to 100 months
  Overall survival (OS)
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival (assessed by the investigators based on RECIST v1.1)
ORR | through study completion, an average of 1 year
  Objective response rate (assessed by independent radiological review and the investigators based on RECIST v1.1))
Duration of response | from the date when CR or PR (whichever recorded earlier) is firstly achieved until the date when disease progression or death is firstly recorded (whichever occurs earlier),assessed up to 2 years
  Duration of response
DCR | the proportion of patients with the best overall response of CR, PR, or stable disease (SD) persisting for 12 weeks
  Disease control rate
PFS2 | From date of randomization until the date of the second documented PD as assessed by the investigator or date of death from any cause, whichever came first, assessed up to 100 months
  Progression-free survival in the next line of treatment(assessed by the investigators based on RECIST v1.1)

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, Study Chair — Center for Cancer Prevention and Treatment of Sun Yat-sen University
Locations (5):
- China (4):
  - Center for Cancer Prevention and Treatment of Sun Yat-sen University, Guangzhou, Guangdong
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Linyi Cancer Hospital, Linyi
  - Fudan University Affiliated Oncology Hospital, Shanghai
- National Cancer Center, Kashiwa, Japan

REFERENCES:
- [Derived] Wang ZX, Peng J, Liang X, Cheng Y, Deng Y, Chen K, Zhang M, Zhang J, Wang W, Cao B, Jin Y, Sun M, Lin Y, Luo S, Li Z, Yang L, Ke Y, Yu H, Li J, Wang Q, Zhu J, Wang F, Xu RH. First-line serplulimab in metastatic colorectal cancer: Phase 2 results of a randomized, double-blind, phase 2/3 trial. Med. 2024 Sep 13;5(9):1150-1163.e3. doi: 10.1016/j.medj.2024.05.009. Epub 2024 Jun 12. PMID 38870931